CLINICAL TRIAL: NCT04315129
Title: Smart Catheter: A Novel Biosensor for Early Detection of Catheter Associated Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17SM4299
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Catheter-Associated Urinary Tract Infection
Keywords: Biosensor

STUDY DESIGN:
Intervention Model Description: Singlearm blinded study in which biosensor diagnosed infection (experiment) will be compared to clinical diagnosis (control) in a single cohort of surgical patients
Masking Description: The biosensors will monitor for infections. As this is an unverified, experimental diagnosis, this will not be made available to the patient or care provider. similarly this will not be available to the clinical researchers in order to avoid observation bias. While the participants, providers and investigators will all be aware that the participants have an active biosensor, they will be blinded to the output thereof.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): A single arm will have biosensor (experimental) diagnoses compared to clinical (control, current standard of care). All participants in this group willl have a biosensor, with the data masked to patients, providers and clinical researchers
  Interventions: Diagnostic Test: Smart Catheter Biosensor

INTERVENTIONS:
Diagnostic Test: Smart Catheter Biosensor — A novel biosensor in-built into the catheter drainage system that monitors the chemical composition of the urine, with the intention of providing early diagnosis of developing infection

SUMMARY:
Urinary Tract Infection (UTI) is the most common hospital acquired infection worldwide, and is most commonly associated with catheterisation of the bladder. Catheter associated urinary tract infection (CAUTI) causes increased hospital costs, increased length of stay and increased mortality. This burden of disease is, in part, mediated by a lack of diagnostic and monitoring modalities for CAUTI. Both traditional and novel UTI diagnostic tests are susceptible to false positives associated with bacterial colonisation, and correlate poorly with clinically meaningful symptomatic CAUTI. As such, the current standard of care is reliant on clinical monitoring, which is susceptible to diagnostic delays, over and under treatment.

Imperial College London have developed a wireless biosensor for continuous monitoring of catheter-urine biochemistry. This project aims to validate this biosensor and demonstrate it's potential for preemptive CAUTI diagnosis through continuous urinary biochemical monitoring.

DETAILED DESCRIPTION:
This research project aims to demonstrate that continuous urinary biochemical monitoring using a Smart Catheter biosensor can provide rapid diagnosis of impending catheter associated urinary tract infection (CAUTI). The primary research question will then be: "Does the Smart Catheter device reduce the time to diagnosis of CAUTI?"

This will be accomplished through four studies: The aim of the first study will be to show the reliability and robustness of the Smart Catheter device through the question: "Is there any difference between the biochemical measurements from the Smart catheter device and a gold-standard laboratory measurement?"

The aim of the second and third studies aim to demonstrate the different biochemical profiles of infected and healthy urine by addressing the research question: "What is the difference in biochemical concentrations in healthy urine as compared to infected urine?" Study 3 will accomplish this by comparing infected human catheter-acquired urine as compared to uninfected human catheter-urine. Study 3 will monitor the changes in biochemical changes in an artifical bladder with artificial urine over time while an infection is induced.

The final study will demonstrate the reduced time to diagnosis in a clinical setting by addressing the research question: " What is the time difference in diagnosis of CAUTI from the CAUTI as compared to the current standard of clinical monitoring?"

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older Subjects expected to undergo catheterisation as part of their clinical care. Signed informed consent is a prerequisite for inclusion in the study.

Exclusion Criteria:

* Consent to participate not given Known sensitivity to urinary catheters or electronic products Patients undergoing urologic procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Time difference of diagnosis | From the time of catheterisation, until 72hours post-removal of catheters.
  The time difference of biosensor diagnosis of catheter associated UTI as compared to clinical diagnosis (defined as the prescription time of new antimicrobials for suspected UTI)

SECONDARY OUTCOMES:
Sensitivity | From the time of catheterisation, until 72hours post-removal of catheters.
  The proportion of those subjects who went on to develop CAUTI did the Smart Catheter correctly predict would have CAUTI?
Specificity | From the time of catheterisation, until 72hours post-removal of catheters.
  The proportion of those subjects who did not go on to develop CAUTI did the Smart Catheter correctly predict would not have CAUTI.
False Positive Rate | From the time of catheterisation, until 72hours post-removal of catheters.
  The proportion of those subjects who would not go on to have CAUTI did the Smart Catheter incorrectly predict would have CAUTI?
False Negative Rate | From the time of catheterisation, until 72hours post-removal of catheters.
  The proportion of those subjects who would go on to have CAUTI did the Smart Catheter incorrectly predict would not have CAUTI?

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital, London, Greater LOndon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant Data is confidential and will to be shared